CLINICAL TRIAL: NCT04111497
Title: A Single-Arm, Open-Label, Phase I/II Study of Glasdegib for Sclerotic Chronic Graft-Vs-Host Disease
Brief Title: Glasdegib for Chronic Graft-Versus-Host Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study closed to accrual early due to side effects of study drug.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Stephanie Lee, Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1005365; NCI-2019-03244 (Registry Identifier: NCI / CTRP); 8771 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Chronic Graft Versus Host Disease; Fasciitis
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Fasciitis | interventions — glasdegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (glasdegib) (Experimental): Patients receive glasdegib PO QD on days 1-28. Cycles repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Glasdegib

INTERVENTIONS:
Drug: Glasdegib — Given PO
  Other Names: 1095173-27-5; PF 04449913; PF-04449913; PF04449913

SUMMARY:
This phase I/II trial studies whether glasdegib is helpful in treating sclerosis associated with chronic graft-versus-host disease. It will also investigate the safety of glasdegib in treating patients with chronic graft-versus-host disease.

DETAILED DESCRIPTION:
OUTLINE: This is a phase I/II study.

Patients receive glasdegib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with moderate or severe cGVHD according to the 2014 National Institute of Health (NIH) Consensus Criteria
* Diagnosed with cGVHD-related sclerosis or fasciitis

  * Skin feature score of at least 2 OR
  * Joints and fascia score of at least 1
* New, stable or progressive sclerosis/fasciitis despite treatment with at least one prior line of systemic therapy for cGVHD
* Female patients who:

  * Are documented to be postmenopausal or are surgically sterile, OR
  * If of childbearing potential, agree to use at least 1 highly effective method of contraception from the time of signing the informed consent form through 30 days after the last dose of study drug, OR agree to practice true abstinence or exclusively non-heterosexual activity when this is in line with the preferred and usual lifestyle of the subject
* Male patients who:

  * Are surgically sterile (vasectomized) OR
  * Agree to use at least 1 highly effective method of contraception during the entire study treatment period and through 30 days after the last dose of study drug, OR agree to practice true abstinence or exclusively non-heterosexual activity when this is in line with the preferred and usual lifestyle of the subject, AND
  * Agree to use a condom to prevent potential transmission of investigational drug in seminal fluid
* Absolute neutrophil count (ANC) > 1000/uL
* Platelet count > 50 x 10^9/mL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2 x upper limit of normal (ULN) unless attributed to cGVHD
* Normal total bilirubin unless attributed to cGVHD
* Creatinine < 2.0 mg/dl

Exclusion Criteria:

* Hospitalization for evaluation or management of an infection within the last 8 weeks
* Known organ dysfunction

  * Uncontrolled cardiovascular disease, including arrhythmias, congestive heart failure
  * Oxygen requirement
* Addition of any new systemic immunosuppressive treatment within the last 2 weeks

  * Addition of new systemic immunosuppressive treatment along with glasdegib is also prohibited
* Corrected QT (QTc) interval > 480 ms
* Female patients who are lactating or have a positive serum pregnancy test
* Major surgery within 14 days before enrollment

  * Does not include placement of venous access device, bone marrow biopsy, GVHD diagnostic biopsy, or other routine procedures in chronic GVHD or post-transplantation care
* Use of any concomitant medications meds that are prohibited within the past 7 days
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known intolerance to glasdegib, sonidegib, or vismodegib
* Non-hematologic malignancy within the past 2 years with the exception of:

  * Adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer
  * Carcinoma in situ of the cervix or breast
  * Prostate cancer of Gleason grade 6 or less with stable prostate-specific antigen levels
  * Cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study
* Treatment with non-Food and Drug Administration (FDA) approved drug within 21 days of start of this trial
* Evidence of recurrent or progressive underlying malignant disease
* Karnofsky performance status < 70%
* History of non-compliance
* Life expectancy < 6 months
* Grade 2 or 3 muscle cramping, or grade 1 muscle cramping that occurs at least weekly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Duke University Medical Center, Durham, North Carolina
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potentially eligible patients were approached at participating study centers during clinic visits.
Pre-assignment Details: After the participant signed and dated the Informed Consent Form (ICF), screening began. Once all screening procedures were completed and eligibility was confirmed, the participant was enrolled into the study. The screening period lasted from the date the participant signed consent until they completed the enrollment visit and started study drug.
Period: Overall Study
Arm/Group | Treatment (Glasdegib)
Started | 15
Completed (Completed means a participant finished study drug per protocol.) | 1
Not Completed | 14
Not completed — relapse of primary disease | 1
Not completed — toxicity and/or lack of efficacy | 13

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Glasdegib)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 64.0 [33 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: Safety assessments will consist of monitoring and recording adverse events.
Time Frame: From the start of treatment through 28 days after stopping study drug (Up to 25 months total)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glasdegib)
Number analyzed (Participants) | 15
Participants
  Participants with an SAE and a non-serious AE | 3
  Participants with a non-serious AE only | 6
  Participants without any adverse events | 6

2. Secondary Outcome: Overall Response Rate (ORR) in Sclerotic Manifestations
Description: ORR will be calculated according to (1) the response definitions of the National Institute of Health (NIH) Consensus Conference for (a) skin or joint scores (0-3), where improvement by at least 1 point is a partial response (PR) and return to score 0 is a complete response (CR), or (b) the photographic range of motion scale (0-25) where improvement by at least 1 point is a PR and return to score 25 is a CR; and (2) change in the 0-10 sclerotic severity scale where at least a 2 point improvement is a PR or return to 0 (CR). Non-responders are those with mixed response (improvement in one regard and worsening in another), unchanged (stable), and progression.
Time Frame: Up to 12 months after starting glasdegib
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glasdegib)
Number analyzed (Participants) | 15
Participants
  Partial response | 7
  Mixed response | 1
  Unchanged | 6
  Progressive | 1

3. Secondary Outcome: ORR in All Chronic Graft Versus Host Disease (cGVHD) Manifestations
Description: ORR will be calculated according to the response definitions of the NIH Consensus Conference.
Time Frame: Up to 12 months after the starting glasdegib
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glasdegib)
Number analyzed (Participants) | 15
Participants
  ORR for all manifestations of chronic GVHD: partial response | 8
  ORR for all manifestations of chronic GVHD: mixed response | 1
  ORR for all manifestations of chronic GVHD: unchanged | 5
  ORR for all manifestations of chronic GVHD: progressive | 1
  ORR for sclerotic manifestations: partial response | 8
  ORR for sclerotic manifestations: mixed response | 1
  ORR for sclerotic manifestations: unchanged | 5
  ORR for sclerotic manifestations: progressive | 1

4. Secondary Outcome: Failure-free Survival
Description: Failure-free survival will be estimated using the Kaplan-Meier method (product limit estimator), with death, relapse, or start of another systemic immunosuppressive agent considered as events. Patients lost to follow-up or who withdraw consent will be censored.
Time Frame: At 12 months
Population: Five patients censored because they left the study before month 12
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Treatment (Glasdegib)
Number analyzed (Participants) | 15
percentage | 37 [10 to 64]

5. Secondary Outcome: Symptom Burden Assessment - Absolute Change
Description: Subjects will provide assessments of their symptom burden using a validated instrument recommended by the NIH Consensus on Chronic GVHD (Lee Chronic GVHD Symptom Scale). These will be collected before starting glasdegib on day 1 of cycle 1, and again on day (D)1, cycles 4, 7, 10 and end of treatment. Summary scores will be calculated based on published algorithms with absolute changes from baseline and clinically meaningful changes described for the population as a whole and based on CR+PR versus (vs.) stable disease (SD)+mixed response (MR)+progressive disease (PD), when adequate data are available for analysis.
  Lee Symptom Scale: minimum 0, maximum 100; higher score is worse outcome.
  Due to lack of adequate data at cycles 7 and 10, only Cycle 4 and End of Treatment are presented
Time Frame: Cycle 4 (day 85) and End of Treatment (up through 24 months) [Due to lack of adequate data at cycles 7 (day 169) and 10 (day 253), they are not presented.]
Population: Data not available for 5 and 4 participants for the Cycle 4 and End of Treatment visits, respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treatment (Glasdegib), All: Patients receive glasdegib PO QD on days 1-28. Cycles repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Glasdegib: Given PO
- CR+PR: Responders (Complete and Partial Response)
- MR+SD+PD: Non-responders (Mixed Response, Stable Disease, and Progressive Disease)
Arm/Group | Treatment (Glasdegib), All | CR+PR | MR+SD+PD
Number analyzed (Participants) | 11 | 7 | 4
score on a scale
  Cycle 4 (Day 85): number analyzed (Participants) | 10 | 7 | 3
  Cycle 4 (Day 85) | 2.5 (6.9) | 4.9 (6.9) | -3.0 (1.5)
  End of Treatment | 2.8 (9.9) | 6.8 (10.5) | -4.1 (1.8)

6. Secondary Outcome: Quality of Life Assessment
Description: Subjects will provide assessments of their quality of life using the NIH-endorsed Patient Reported Outcomes Measurement Information System (PROMIS)-29. These will be collected before starting glasdegib on day 1 of cycle 1, and again on day (D)1, cycles 4, 7, 10 and end of treatment. Scores will be calculated based on published algorithms with absolute changes from baseline for the population as a whole and based on CR+PR versus stable disease (SD)+mixed response (MR)+progressive disease (PD), when adequate data are available for analysis.
  PROMIS-29 theoretical minimums and maximums are as follows:
  Physical Function: 22.5-57.0 Depression: 41.0-79.4 Anxiety: 40.3-81.6 Sleep Disturbance: 32.0-73.3 Fatigue: 33.7-75.8 Ability to Participate in Social Roles: 27.5-64.2 Pain Interference: 41.6-75.6 Higher score means a better outcome for Physical Function, Sleep Disturbance, and Social Roles.
  Higher score means a worse outcome for Anxiety, Depression, Fatigue, and Pain Interference.
Time Frame: Cycle 4 (day 85) and End of Treatment (up through 24 months) [Due to lack of adequate data at cycles 7 (day 169) and 10 (day 253) they are not presented.]
Population: Data not available for 5 participants at Cycle 4 and 4 participants for End of Treatment (EOT)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment (Glasdegib), All | CR+PR | MR+SD+PD
Number analyzed (Participants) | 11 | 7 | 4
score on a scale
  Cycle 4 (day 85) - Physical Function absolute change: number analyzed (Participants) | 10 | 7 | 3
  Cycle 4 (day 85) - Physical Function absolute change | 0.3 (5.2) | 0.8 (6.2) | -0.9 (2.2)
  Cycle 4 (day 85) - Anxiety absolute change: number analyzed (Participants) | 11 | 7 | 3
  Cycle 4 (day 85) - Anxiety absolute change | 2.1 (5.9) | 1.6 (6.8) | 3.4 (3.9)
  Cycle 4 (day 85) - Depression absolute change: number analyzed (Participants) | 11 | 7 | 3
  Cycle 4 (day 85) - Depression absolute change | 0.3 (8.2) | -0.6 (9.6) | 2.2 (3.9)
  Cycle 4 (day 85) - Fatigue absolute change: number analyzed (Participants) | 11 | 7 | 3
  Cycle 4 (day 85) - Fatigue absolute change | -0.4 (6.8) | -2.7 (6.7) | 4.9 (3.7)
  Cycle 4 (day 85) - Sleep Disturbance absolute change: number analyzed (Participants) | 11 | 7 | 3
  Cycle 4 (day 85) - Sleep Disturbance absolute change | 0.5 (5.5) | 1.4 (5.8) | -1.6 (5.0)
  Cycle 4 (day 85) - Ability to Participate in Social Roles absolute change: number analyzed (Participants) | 11 | 7 | 3
  Cycle 4 (day 85) - Ability to Participate in Social Roles absolute change | 2.1 (7.4) | 2.7 (8.9) | 0.6 (2.8)
  Cycle 4 (day 85) - Pain Interference absolute change: number analyzed (Participants) | 11 | 7 | 3
  Cycle 4 (day 85) - Pain Interference absolute change | -1.8 (9.9) | -5.8 (7.7) | 7.6 (8.7)
  End of Treatment - Physical Function absolute change | -0.1 (4.9) | -0.1 (6.0) | 0.1 (2.5)
  End of Treatment - Anxiety absolute change | 0.8 (5.3) | 2.5 (4.4) | -2.1 (6.0)
  End of Treatment - Depression absolute change | 0.2 (5.0) | -0.2 (5.7) | 1.0 (4.0)
  End of Treatment - Fatigue absolute change | -1.7 (5.1) | -0.7 (4.1) | -3.5 (6.8)
  End of Treatment - Sleep Disturbance absolute change | 1.3 (5.0) | 0.3 (4.1) | 2.9 (6.7)
  End of Treatment - Ability to Participate in Social Roles absolute change | -0.5 (5.1) | -2.3 (5.5) | 2.7 (2.0)
  End of Treatment - Pain Interference absolute change: number analyzed (Participants) | 10 | 7 | 4
  End of Treatment - Pain Interference absolute change | 3.1 (8.7) | 2.4 (9.2) | 4.4 (9.0)

7. Secondary Outcome: Biologic Impact of Hedgehog Pathway Inhibition
Description: Banking of blood and skin biopsy material for future biologic studies of hedgehog pathway inhibition.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glasdegib)
Number analyzed (Participants) | 15
Participants | 15

8. Secondary Outcome: Symptom Burden Assessment - Clinically Meaningful Change
Description: as for outcome 5
Time Frame: as for outcome 5
Population: Data not available for 5 and 4 participants at the Cycle 4 and End of Treatment (EOT) visits, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glasdegib), All | CR+PR | MR+SD+PD
Number analyzed (Participants) | 11 | 7 | 4
Participants
  Cycle 4 (Day 85): number analyzed (Participants) | 10 | 7 | 3
  Cycle 4 (Day 85): Better | 0 | 0 | 0
  Cycle 4 (Day 85): No change | 6 | 3 | 0
  Cycle 4 (Day 85): Worse | 4 | 4 | 3
  End of Treatment: Better | 2 | 1 | 1
  End of Treatment: No change | 5 | 2 | 3
  End of Treatment: Worse | 4 | 4 | 0

9. Secondary Outcome: Quality of Life Assessment - Clinically Meaningful Change
Description: Subjects will provide assessments of their quality of life using the NIH-endorsed Patient Reported Outcomes Measurement Information System (PROMIS)-29. These will be collected before starting glasdegib on day 1 of cycle 1, and again on day (D)1, cycles 4, 7, 10 and end of treatment. Scores for physical functioning will be calculated based on published algorithms with clinically meaningful changes described for the population as a whole and based on CR+PR versus (vs.) stable disease (SD)+mixed response (MR)+progressive disease (PD), when adequate data are available for analysis.
  PROMIS-29 minimums and maximums as follows:
  Physical Function: 22.5-57.0 Depression: 41.0-79.4 Anxiety: 40.3-81.6 Sleep Disturbance: 32.0-73.3 Fatigue: 33.7-75.8 Ability to Participate in Social Roles: 27.5-64.2 Pain Interference: 41.6-75.6 Higher score means a better outcome for Physical Function, Sleep, and Social Roles.
  Higher score means a worse outcome for Anxiety, Depression, Fatigue, and Pain.
Time Frame: as for outcome 6
Population: Data not available for 5 and 4 participants at the Cycle 4 and End of Treatment (EOT) visits, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glasdegib), All | CR+PR | MR+SD+PD
Number analyzed (Participants) | 11 | 7 | 4
Participants
  Cycle 4 (Day 85) - Physical Function clinically meaningful change: number analyzed (Participants) | 10 | 7 | 3
  Cycle 4 (Day 85) - Physical Function clinically meaningful change: Better | 1 | 1 | 0
  Cycle 4 (Day 85) - Physical Function clinically meaningful change: No change | 8 | 5 | 3
  Cycle 4 (Day 85) - Physical Function clinically meaningful change: Worse | 1 | 1 | 0
  Cycle 4 (Day 85) - Anxiety clinically meaningful change: number analyzed (Participants) | 10 | 7 | 3
  Cycle 4 (Day 85) - Anxiety clinically meaningful change: Better | 1 | 1 | 0
  Cycle 4 (Day 85) - Anxiety clinically meaningful change: No change | 6 | 4 | 2
  Cycle 4 (Day 85) - Anxiety clinically meaningful change: Worse | 3 | 2 | 1
  Cycle 4 (Day 85)- Depression clinically meaningful change: number analyzed (Participants) | 10 | 7 | 3
  Cycle 4 (Day 85)- Depression clinically meaningful change: Better | 2 | 2 | 0
  Cycle 4 (Day 85)- Depression clinically meaningful change: No change | 6 | 4 | 2
  Cycle 4 (Day 85)- Depression clinically meaningful change: Worse | 2 | 1 | 1
  Cycle 4 (Day 85)- Fatigue clinically meaningful change: number analyzed (Participants) | 10 | 7 | 3
  Cycle 4 (Day 85)- Fatigue clinically meaningful change: Better | 1 | 1 | 0
  Cycle 4 (Day 85)- Fatigue clinically meaningful change: No change | 7 | 5 | 2
  Cycle 4 (Day 85)- Fatigue clinically meaningful change: Worse | 2 | 1 | 1
  Cycle 4 (Day 85) - Sleep Disturbance clinically meaningful change: number analyzed (Participants) | 10 | 7 | 3
  Cycle 4 (Day 85) - Sleep Disturbance clinically meaningful change: Better | 2 | 1 | 1
  Cycle 4 (Day 85) - Sleep Disturbance clinically meaningful change: No change | 6 | 4 | 2
  Cycle 4 (Day 85) - Sleep Disturbance clinically meaningful change: Worse | 2 | 2 | 0
  Cycle 4 (Day 85) - Ability to Participate in Social Roles clinically meaningful change: number analyzed (Participants) | 10 | 7 | 3
  Cycle 4 (Day 85) - Ability to Participate in Social Roles clinically meaningful change: Better | 3 | 3 | 0
  Cycle 4 (Day 85) - Ability to Participate in Social Roles clinically meaningful change: No change | 6 | 3 | 3
  Cycle 4 (Day 85) - Ability to Participate in Social Roles clinically meaningful change: Worse | 1 | 1 | 0
  Cycle 4 (Day 85) - Pain Interference clinically meaningful change: number analyzed (Participants) | 10 | 7 | 3
  Cycle 4 (Day 85) - Pain Interference clinically meaningful change: Better | 3 | 3 | 0
  Cycle 4 (Day 85) - Pain Interference clinically meaningful change: No change | 5 | 4 | 1
  Cycle 4 (Day 85) - Pain Interference clinically meaningful change: Worse | 2 | 0 | 2
  End of Treatment - Physical Function clinically meaningful change: Better | 1 | 1 | 0
  End of Treatment - Physical Function clinically meaningful change: No change | 9 | 5 | 4
  End of Treatment - Physical Function clinically meaningful change: Worse | 1 | 1 | 0
  End of Treatment - Anxiety clinically meaningful change: Better | 1 | 0 | 1
  End of Treatment - Anxiety clinically meaningful change: No change | 8 | 5 | 3
  End of Treatment - Anxiety clinically meaningful change: Worse | 2 | 2 | 0
  End of Treatment - Depression clinically meaningful change: Better | 1 | 1 | 0
  End of Treatment - Depression clinically meaningful change: No change | 8 | 5 | 3
  End of Treatment - Depression clinically meaningful change: Worse | 2 | 1 | 1
  End of Treatment - Fatigue clinically meaningful change: Better | 2 | 0 | 2
  End of Treatment - Fatigue clinically meaningful change: No change | 8 | 6 | 2
  End of Treatment - Fatigue clinically meaningful change: Worse | 1 | 1 | 0
  End of Treatment - Sleep Disturbance clinically meaningful change: Better | 2 | 1 | 1
  End of Treatment - Sleep Disturbance clinically meaningful change: No change | 8 | 6 | 2
  End of Treatment - Sleep Disturbance clinically meaningful change: Worse | 1 | 0 | 1
  End of Treatment - Ability to Participate in Social Roles clinically meaningful change: Better | 0 | 0 | 0
  End of Treatment - Ability to Participate in Social Roles clinically meaningful change: No change | 10 | 6 | 4
  End of Treatment - Ability to Participate in Social Roles clinically meaningful change: Worse | 1 | 1 | 0
  End of Treatment - Pain Interference clinically meaningful change: Better | 1 | 1 | 0
  End of Treatment - Pain Interference clinically meaningful change: No change | 7 | 4 | 3
  End of Treatment - Pain Interference clinically meaningful change: Worse | 3 | 2 | 1

ADVERSE EVENTS:
Time Frame: The AE reporting period for this study began when the participant received their first dose of study drug and ended with the EOT visit, or 28 days after the last dose of study drug, whichever was later. Exceptions to this reporting period were (a) any AE occurring due to a protocol-specific screening procedure; and (b) any SAE occuring beyond 28 days after the last dose of glasdegib AND assessed by the investigator as possibly related to glasdegib.
Description: The study collected Grade 3 and above adverse events, with these exceptions:
  An abnormal lab value; unless it led to discontinuation, delay, or modification in treatment, therapeutic intervention, the investigator considered it to be clinically significant, or it met seriousness criteria.
  Chronic GVHD manifestations were not collected as AE's unless they meet seriousness criteria.
  Hospitalization for elective treatment of a stable pre-existing condition was not considered an adverse event.
Arm/Group | Treatment (Glasdegib)
All-Cause Mortality (participants affected / at risk) | 2/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Glasdegib) (N=15)
acute myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) — progressive generalized muscle weakness of unclear etiology, most consistent with acute myopathy
upper respiratory infection (Infections and infestations) | 1 (1) — symptoms suggestive of a URI, increased oxygen needs, no infectious agent identified
mastitis (Infections and infestations) | 1 (1) — infected breast wound of unclear etiology
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Glasdegib) (N=15)
muscle cramping (Musculoskeletal and connective tissue disorders) | 5 (5)
hyponatremia (Metabolism and nutrition disorders) | 2 (2)
hypokalemia (Metabolism and nutrition disorders) | 2 (2)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination led to a smaller than planned number of participants. Several participants met a study-defined endpoint (e.g. starting a new systemic GVHD therapy) or withdrew from the study after stopping study drug, limiting our ability to assess patient-reported outcomes over the long term.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT04111497/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT04111497/ICF_002.pdf